CLINICAL TRIAL: NCT01299493
Title: Systems Intervention to Promote Colorectal Cancer Screening/ Program for the Elimination of Cancer Disparities
Brief Title: Systems Intervention to Promote Colorectal Cancer (CRC) Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 10-1131 / 201110005; U54CA153460 (NIH)
Record Dates: First submitted 2011-02-16; First posted 2011-02-18 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Carcinoma
Keywords: carcinoma; colorectal cancer; community health centers; cluster-randomized; health behavior
MeSH Terms: conditions — Carcinoma; Colorectal Neoplasms; Health Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): Access to systems-level interventions to increase colorectal cancer screening.
  Interventions: Other: Systems-level intervention to promote colon cancer screening
- Usual Care (No Intervention): Practices will receive access to intervention components after outcomes data collection is complete.

INTERVENTIONS:
Other: Systems-level intervention to promote colon cancer screening — Intervention practices will receive access to, and assistance in implementing, evidence-based strategies for increasing colorectal cancer screening rates.
  Arms: Interventional

SUMMARY:
Colorectal cancer is the second leading cause of cancer death and one of the most commonly diagnosed malignancies. Screening is effective at reducing incidence and mortality from colorectal cancer. This study will evaluate the effectiveness of implementing systems-changes in community health centers that facilitate screening.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is one of the cancers that our community partners have identified as a priority. It is the second leading cause of cancer death in the United States, and one with significant disparities in screening, stage of diagnosis, and survival. Underinsured and uninsured adults are less likely to be screened, more likely to have their cancer diagnosed at a late stage, and less likely to survive CRC. In this project we will work with "safety-net" health centers serving Medicaid and uninsured patients in St. Louis City and St. Louis County in Missouri, and in East St. Louis/St. Clair County in Illinois. Working with our Colorectal Cancer Community Partnership we planned a cluster-randomized delayed start trial to test the effectiveness of offering community health centers a "Menu" of evidence-based systems interventions for increasing rates of CRC screening. The strategies included in the Menu will be drawn from evidence-based interventions. The control condition will be usual care, but in concordance with our partners' wishes, we will offer all participating health centers access to state-of-the-art evidence-based patient education materials. The primary outcome will be CRC screening adherence as measured by self-report surveys of a random sample of health center patients. Our evaluation will also be informed by a chart audit to assess screening referral and completion, surveys of physicians and staff at intervention sites to assess implementation outcomes, and exit interviews with administration of intervention health centers to assess maintenance of the intervention strategies. We developed and will conduct our study adhering to the principles of community-based participatory research (CBPR). The specific aims are: (1) Working with community partners, we will select and refine the evidence-based intervention strategies for the trial; (2) Using a CBPR approach, we will collaborate with our partners to implement and evaluate the systems-level intervention for its effectiveness in increasing CRC screening rates. (3) Using the RE-AIM framework, we will work with our partners to evaluate implementation and maintenance of systems changes by intervention health centers and adoption of the changes by control centers. Compared to traditional clinics and healthcare providers, safety-net health centers face additional challenges in implementing evidence-based strategies for increase screening uptake; yet rigorously testing such strategies in this context is novel. Allowing health centers to select from a menu of strategies will provide a practical test of effectiveness, and will increase buy-in and representativeness of participating health centers. As a practical clinical trial with good external validity, this project has the potential for significant impact on CRC screening rates with promise for substantial impact on disparities in CRC burden. This study is responsive to community concerns about CRC and about no-intervention control groups, and is responsive to the RFA by proposing a CBPR randomized controlled trial to increase access to and utilization of CRC screening procedures.

ELIGIBILITY:
Inclusion Criteria:

* Community health center in the Saint Louis Metropolitan Area, including Southern Illinois
* Participant in Partnership Planning Process
* Affiliated with the Washington University Program for the Elimination of Cancer Disparities

Exclusion Criteria:

* Primary patient population has private health insurance.
* Not in an medically underserved area.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2012-06-19 (Actual); Primary Completion 2017-09-21 (Actual); Study Completion 2017-09-21 (Actual)

PRIMARY OUTCOMES:
Practice-level colon cancer screening rate | 12-months post baseline
  Colorectal cancer screening will be assessed as the proportion of screening-eligible patients who are adherent to national screening guidelines for colorectal cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Aimee S James, PhD, MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] James AS, Richardson V, Wang JS, Proctor EK, Colditz GA. Systems intervention to promote colon cancer screening in safety net settings: protocol for a community-based participatory randomized controlled trial. Implement Sci. 2013 Jun 3;8:58. doi: 10.1186/1748-5908-8-58. PMID 23731594
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu